CLINICAL TRIAL: NCT00044577
Title: See Detailed Description
Brief Title: New Tablet Containing Two FDA Approved Anti-HIV Drugs For Antiretroviral Therapy Experienced HIV-1 Infected Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAL30001
Record Dates: First submitted 2002-08-30; First posted 2002-09-04 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV Infection
Keywords: HIV-1 Abacavir Lamivudine Tenofovir
MeSH Terms: conditions — Infections; HIV Infections | interventions — abacavir, lamivudine drug combination; abacavir; Lamivudine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: abacavir/lamivudine
Drug: abacavir
Drug: lamivudine
Drug: tenofovir
  Other Names: lamivudine; abacavir/lamivudine; abacavir

SUMMARY:
A 48-week study to investigate the safety and effectiveness of a new compact formulation of two already FDA-approved anti-HIV drugs in subjects who have already been receiving treatment for their HIV infection.

DETAILED DESCRIPTION:
A phase III, randomized, open-label, parallel, multicenter study to evaluate treatment with fixed-dose combination of abacavir/lamivudine (600mg/300mg) once-daily versus abacavir (300mg) twice-daily and lamivudine (300mg) once-daily in combination with tenofovir once-daily and a new PI or NNRTI for 48 weeks in ART-experienced HIV-1 infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Antiretroviral therapy (ART) experienced and currently receiving a stable regimen containing 3 nucleoside reverse transcriptase inhibitors (NRTIs), or 2 NRTIs plus a protease inhibitor (PI) or non-nucleoside reverse transcriptase inhibitors (NNRTI) for at least 3 months (there should be no significant ART modifications for at least 3 months and no ART change anticipated between Screening and initiation of the study therapy).
* Patients must be naive to tenofovir.
* HIV-1 RNA level > 1000 copies/ml on at least one occasion within 21 days of study entry.
* A CD4 cell count > 50 cells/mm3.
* Specified viral genotypes.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Has an active diagnosis of AIDS.
* Additional qualifying criteria to be determined by the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166
Dates: Start 2002-07-16 (Actual); Primary Completion 2004-05-25 (Actual); Study Completion 2004-05-25 (Actual)

PRIMARY OUTCOMES:
HIV viral load response as measured by change from baseline in HIV-1 RNA over 24 and 48 weeks. Safety | 48 weeks

SECONDARY OUTCOMES:
Viral load response T-cell count Health Outcomes Resistance

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (58):
- United States (23):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Seattle, Washington
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Canada (5):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- France (5):
  - GSK Investigational Site, Garches
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Levallois-Perret
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
- Germany (4):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Hamburg
- Italy (6):
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Verona, Veneto
- Portugal (5):
  - GSK Investigational Site, Braga
  - GSK Investigational Site, Cascais
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Faro
  - GSK Investigational Site, Lisbon
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
- United Kingdom (3):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Thornton Heath, Surrey
  - GSK Investigational Site, London

REFERENCES:
- [Result] EFFICACY AND SAFETY OF A ONCE DAILY FIXED-DOSE COMBINATION OF ABACAVIR/LAMIVUDINE (ABC/3TC) [FDC ] VERSUS ABC TWICE DAILY AND 3TC ONCE DAILY AS SEPARATE ENTITIES [SE] IN ART-EXPERIENCED HIV-1 INFECTED SUBJECTS (CAL30001): 48 WEEK DATA. Clumeck, N., LaMarca, A., Fu, K., Gordon, D., Craig, C., Zhao, H. , Paes, D., and Scott, T. (WePe6.3C13), 3rd International AIDS Society Conference on HIV Pathogenesis and Treatment, Rio de Janeiro; Brazil, 7/24/2005
- [Result] C Craig, C Stone, T Bonny, K Fu. Similar virology findings in ABC/3TC fixed dose combination (FDC) OAD compared with standard dosing in experienced subjects (CAL30001, ALTO). 7th ICDTHI, Glasgow, UK, 14-18 November 2004. Abstract 98
- [Result] Clumeck N, Lamarca A, Fu K, Gordon D, Craig C, Zhao H, Paes D, Scott T. Safety and efficacy of a once daily (OAD) Fixed-Dose Combination (FDC) of ABC/3TC [FDC arm] versus ABC twice daily (BID) and 3TC OAD as separate entities [SE arm] in ART-Experienced HIV-1 Infected Patients. 44th ICAAC, Washington, DC, 30 October-2 November 2004. Abstr. H-558